CLINICAL TRIAL: NCT02292472
Title: A Randomized, Double-blind, Multi-center, Phase II Optimal Dose-finding Study to Determine Safety and Efficacy of Medytoxin® in Subjects in Benign Masseteric Hypertrophy
Brief Title: Medytoxin® Treatment in Patients With Benign Masseteric Hypertrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT_PRT_BMH01
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Hypertrophy of Masseter Muscle
Keywords: masticatory muscles
MeSH Terms: conditions — Masticatory Muscles, Hypertrophy of | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medytoxin® (Experimental): Botulinum toxin type A
  Interventions: Drug: Botulinum Toxin Type A
- Normal Saline (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Inject intramuscularly once in visit 2
  Other Names: Medytoxin®
  Arms: Medytoxin®
Drug: Placebos — Inject intramuscularly once in visit 2
  Other Names: Normal saline
  Arms: Normal Saline

SUMMARY:
This study design is A Randomized, Double-blind, Multi-center, Phase II Optimal Dose-finding Study to Determine the Safety and Efficacy of Meditoxin® in Subjects in Benign Masseteric Hypertrophy.

DETAILED DESCRIPTION:
Subjects who voluntarily signed the informed consent and are judged to be eligible for this study will be intramuscularly injected with the study drug or the placebo to find appropreate dose for the treatment of Benign Masseteric Hypertrophy. Thereafter, follow-up visits will be made and efficacy and safety assessment will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who shows benign masseteric hypertrophy
2. Male or female subject over 19 years of age and written informed consent is obtained from the patient or LAR.
3. Subject who has bisymmetry of masster at visual assessment.
4. Subejects who qualifies the standard meets on ultrasonics wave value.
5. Subjects who can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. Diagnosis of myasthenia, facial palsy or severe facial asymmetry
2. Subject who got any treatment, including double jaw surgery, laser, thread treatment etc. in 1 year.
3. Subject who had previously received botulinum toxin within 3 months prior to the study entry
4. Subject who is participating in other investigational study at present or 30 prior to the screening date.
5. Subject with known hypersensitivity to botulinum toxin
6. Subject who are pregnant or lactating or found pregnancy though the urine or sebum test or disagreed to avoid pregnancy during study preiod.
7. Subjects who are not eligible for this study at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2015-05-24 (Actual); Study Completion 2015-08-24 (Actual)

PRIMARY OUTCOMES:
Reduction amount of masseter muscle thickness | after the injection

SECONDARY OUTCOMES:
Reduction amount of masseter muscle thickness and lower face volume | after the injection
Overall satisfaction of subject | after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, Ph D, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chungang university hospital, Seoul, South Korea